CLINICAL TRIAL: NCT05902754
Title: Broccoli Extract Supplementation and Gastrointestinal Health in Older Adults With Active Alcohol Use and Low Diet Quality
Brief Title: Broccoli Extract Supplementation in Older Adults With Alcohol Use Disorder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Aline Zaparte, Principal Investigator, Louisiana State University Health Sciences Center in New Orleans
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 1268; U24DK132740 (NIH)
Record Dates: First submitted 2023-05-25; First posted 2023-06-15 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Alcohol Use Disorder
Keywords: Inflammation; Leaky gut; Supplements
MeSH Terms: conditions — Alcoholism; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Labels of the product will be replaced with "Tablets A" and "Tablets B" labels.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sulforaphane tablets (Experimental): People in the experimental group will be advised to take 2 tablets a day with a meal for 28 days.
  Interventions: Dietary Supplement: Generally Recognized as Safe - Sulforaphane
- Placebo tablets (Placebo Comparator): People in the placebo group will be advised to take 2 tablets a day with a meal for 28 days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Generally Recognized as Safe - Sulforaphane — Participants will be asked to maintain the same food ingestion habits as before the study and take 2 tablets of Sulforaphane a day with a meal for 28 days.
  Other Names: Avmacol
  Arms: Sulforaphane tablets
Dietary Supplement: Placebo — Participants will be asked to maintain the same food ingestion habits as before the study and take 2 tablets of placebo a day with a meal for 28 days.
  Other Names: Inactive tablets
  Arms: Placebo tablets

SUMMARY:
Chronic alcohol consumption leads to perturbations in gut microbiome balance (dysbiosis) and disruption of gut barrier integrity. As a result, bacteria, toxins, and metabolites can enter the blood stream and reach distant organs, triggering inflammation and oxidative stress. Through this mechanism gut leak is closely related to the onset of metabolic diseases, such as nonalcoholic fatty liver disease (NAFLD) and diabetes.

Despite the prominent role of diet and alcohol in the pathogenesis of metabolic diseases, there is a lack of treatments to mitigate their effects in triggering systemic inflammation and oxidative stress. Novel treatments using generally recognized as safe (GRAS) compounds focused on restoring the intestinal barrier to mitigate metabolite endotoxemia are sorely needed. This project will test the potential of broccoli sprouts extract (BSE) as a GRAS treatment to minimize the combined effect of poor nutrition and alcohol on the gut. Broccoli sprouts are rich in sulforaphane, a bioactive compound derived from the glucosinolate glucoraphanin with anti-inflammatory and antioxidant proprieties. BSE supplementation has been used in preclinical and clinical studies as a health- promoting food, showing significant positive changes in the gut microbiota composition, protection against colitis, cardiometabolic improvement, and lower inflammation. We believe that BSE is a viable alternative therapeutic approach for patients who are resistant to lifestyle changes such as healthy eating and reducing alcohol use. Our purpose is to test BSE supplementation in human subjects with poor nutrition compounded by alcohol use, specifically in older adults who we believe will receive greater benefit from this approach. At the completion of the proposed study, we expect to have determined that treatments using generally recognized as safe (GRAS) compounds can be useful to restore the gut barrier integrity, and as consequence of reduced gut leak we expect to observe lower inflammation and oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥ 50 years of age at enrollment.
* Consume at least 8 alcoholic drinks/week. AUDIT-C score >8.

Exclusion Criteria:

* Bowel-related diseases
* Diagnosed Diabetes
* Allergy or intolerance to broccoli.
* Any acute illness within the last 6 weeks.
* Chronic anti-inflammatory use or antibiotic treatment in the last 7 days.
* Acute illness within the preceding six weeks (defined as fever, new antibiotic use or unscheduled healthcare visit - for illness).
* Acute alcohol intoxication upon arrival on the day of study visit.

Additional exclusion criteria:

• Any health issue that, the study investigator's judgement, confers excess risk for participation.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2024-12-08 (Actual); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Change on the Leaky gut biomarker | Change in serum levels of intestine acid biding proteins after 28 days of intervention.
  Measured by serum levels of intestine acid biding proteins.
Change of Inflammation biomarkers | Change in serum Interleukin-6 levels after 28 days of intervention.
  Measured by serum Interleukin-6 level.

CONTACTS AND LOCATIONS:
Overall Officials: Aline Zaparte, PhD, Principal Investigator — Postdoctoral Fellow
Locations (1):
- Louisiana Health Sciences Center, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No